CLINICAL TRIAL: NCT04796831
Title: An Open Label Study to Determine the Absolute Oral Bioavailability of Quizartinib Using a Radiolabeled Microtracer in Healthy Subjects
Brief Title: A Study to Determine the Absolute Oral Bioavailability of Quizartinib Using a Radiolabeled Microtracer in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-U107; 2021-000198-10 (EudraCT Number)
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-04

CONDITIONS: Healthy Subjects
Keywords: Quizartinib; Healthy Subjects; Pharmacokinetics; Oral Bioavailability; Microtracer
MeSH Terms: interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Participants who will receive a single, oral dose of 60 mg quizartinib and a single, IV administration of 50 μg 14C-quizartinib solution for infusion at 4 hours post-oral dosing.
  Interventions: Drug: Quizartinib dihydrochloride; Drug: 14C-Quizartinib solution for infusion

INTERVENTIONS:
Drug: Quizartinib dihydrochloride — Single oral dose of 60 mg quizartinib (2 x 30 mg tablets)
  Other Names: Quizartinib
Drug: 14C-Quizartinib solution for infusion — 50 μg solution for infusion containing NMT 22.84 kBq 14C in 5 mL; administered once as a 15-minute infusion

SUMMARY:
Quizartinib, a selective FLT3 inhibitor, is being developed as a treatment for acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). The absolute oral bioavailability of quizartinib has not yet been studied. This study is designed to estimate quizartinib bioavailability of quizartinib following oral and intravenous (IV) administration.

DETAILED DESCRIPTION:
Quizartinib bioavailability based on the dose-adjusted exposure of quizartinib following oral and IV administration will be assessed in healthy male subjects. The primary objective of this study is to determine the absolute oral bioavailability of quizartinib. Secondary objectives will include characterizing the plasma PK of quizartinib, radiolabeled quizartinib, and the major circulating metabolite after a single oral dose and IV administration. Safety and tolerability of quizartinib will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18 years to 55 years of age (inclusive) at the time of signing informed consent
* Body mass index (BMI) of 18.0 kg/m^2 to 32.0 kg/m^2 (inclusive) at screening

Exclusion Criteria:

* History or presence of:

  * Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease, as judged by the Investigator.
  * Any other condition, including laboratory abnormality, that in the opinion of the Investigator, would jeopardize the safety of the subject, obtaining informed consent, compliance to the study procedures, or the validity of the study results.
* History of a clinically significant illness, in the opinion of the Investigator, within 4 weeks prior to administration of quizartinib.
* History, or presence in the average of triplicate ECGs at screening and admission (Day -1), of any of the following cardiac conduction abnormalities:

  * QT interval corrected with Fridericia's formula (QTcF) > 450 milliseconds (ms).
  * Evidence of second- or third-degree atrioventricular block.
  * Evidence of complete left or right bundle branch block.
  * QRS or T wave morphology that could, in the Investigator's opinion, render QT interval assessment unreliable (confirmed with triplicate ECG).
* Laboratory results (serum chemistry, hematology, coagulation, and urinalysis) outside the normal range, if considered clinically significant by the Investigator at screening or admission (Day -1).
* Estimated creatinine clearance (CrCl) <90 mL/min (calculated using Cockcroft-Gault Equation) at screening.
* Use of drugs with a risk of QT interval prolongation or Torsades de Pointes (TdP) within 14 days of admission (Day -1) (or 5 drug half-lives, if 5 drug half-lives are expected to exceed 14 days).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants who met all inclusion criteria and no exclusion criteria were included in this study and were enrolled at 1 clinic center in the United Kingdom.
Pre-assignment Details: Participants underwent preliminary screening procedures up to 21 days before investigational medicinal product (IMP) administration (Day -21 to Day-2). Participants were admitted in the morning on the day prior to IMP administration (i.e., Day -1), at which time admission procedures were undertaken to confirm eligibility. Participants were dosed in the morning of Day 1 following an overnight fast of a minimum of 8 hours for the oral dose (a minimum of 12 hours for the intravenous dose).
Groups:
- All Participants: Participants who received a single, oral dose of 60 mg quizartinib and a single, IV administration of 50 μg 14C-quizartinib solution for infusion at 4 hours post-oral dosing.
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patient demographic and baseline characteristics were reported from the Safety Population.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Absolute Oral Bioavailability for Quizartinib As Assessed By Pharmacokinetic Parameters for Area Under the Plasma Concentration-Time Curve Following Intravenous and Oral Administrations of Quizartinib
Description: The absolute bioavailability assessment for quizartinib was based on the pharmacokinetic parameters area under the curve (AUC) from the time of dosing to time Tlast (AUClast) and AUC from the time of dosing extrapolated to infinity (AUCinf) for quizartinib following intravenous and oral administrations. Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0).
Time Frame: Relative to oral dosing: Pre-dose and at 1, 2, 4, 4.25, 4.5, 4.75, 5, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, 336, 384, 432, 480, and 504 hours
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: percentage of oral bioavailability
Arm/Group | All Participants
Number analyzed (Participants) | 8
percentage of oral bioavailability
  Area under the concentration-time curve from the time of dosing to time Tlast (AUClast) | 72.12 (7.18)
  Area under the concentration-time curve from the time of dosing extrapolated to infinity (AUCinf) | 71.47 (7.34)

2. Secondary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Plasma Concentration (Cmax) Following Oral Administrations of Quizartinib
Description: Maximum (peak) plasma concentration (Cmax) was an observed value from the study. Cmax was assessed for Quizartinib and active metabolite AC886.
Time Frame: Relative to oral dosing: Pre-dose, 1, 2, 4, 4.25, 4.5, 4.75, 5, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, 336, 384, 432, 480, and 504 hours
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All Participants
Number analyzed (Participants) | 8
ng/mL
  Oral (plasma): Quizartinib | 209 (33.4)
  Oral (plasma): AC886 | 40.7 (24.0)

3. Secondary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Plasma Concentration (Cmax) Following Intravenous Administrations of Quizartinib
Description: Maximum (peak) plasma concentration (Cmax) was an observed value from the study. Cmax was assessed for 14C-Quizartinib and 14C-AC886.
Time Frame: Relative to oral dosing: 4, 4.25, 4.5, 4.75, 5, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, 336, 384, 432, 480, and 504 hours
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 7
pg/mL
  14C-Quizartinib | 1030 (317)
  14C-AC886 | 31.9 (11.4)

4. Secondary Outcome: Pharmacokinetic Parameter of Time to Maximum Plasma Concentration (Tmax) Following Intravenous and Oral Administrations of Quizartinib
Description: Time to maximum plasma concentration (Tmax) was an observed value from the study. Tmax was assessed for Quizartinib and AC886.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Median (Full Range); unit: hours
Arm/Group | All Participants
Number analyzed (Participants) | 8
hours
  Oral (plasma): Quizartinib | 4.75 [2.00 to 5.02]
  Oral (plasma): AC886 | 5.51 [4.75 to 72.12]
  Intravenous: Quizartinib: number analyzed (Participants) | 7
  Intravenous: Quizartinib | 0.25 [0.23 to 0.27]
  Intravenous: AC886: number analyzed (Participants) | 7
  Intravenous: AC886 | 44.02 [20.02 to 68.12]

5. Secondary Outcome: Pharmacokinetic Parameter of Terminal Half-Life (t1/2) Following Intravenous and Oral Administrations of Quizartinib
Description: Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0). Half-life (t1/2) was assessed for Quizartinib, 14C-Quizartinib, AC886, 14C-AC886.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Participants
Number analyzed (Participants) | 8
hours
  Oral (plasma): Quizartinib | 94.2 (23.7)
  Oral (plasma): AC886 | 111 (45.4)
  Intravenous: Quizartinib | 95.7 (29.7)
  Intravenous: AC886: number analyzed (Participants) | 7
  Intravenous: AC886 | 90.4 (31.2)

6. Secondary Outcome: Pharmacokinetic Parameter for Area Under the Plasma Concentration-Time Curve (AUC) Following Oral Administrations of Quizartinib
Description: Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0). Area under the concentration-time curve from the time of dosing to time (AUClast) and area under the concentration-time curve from the time of dosing extrapolated to infinity (AUCinf) were assessed for Quizartinib and AC886.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | All Participants
Number analyzed (Participants) | 8
ng*h/mL
  Oral (plasma): Quizartinib, AUClast | 17000 (4990)
  Oral (plasma): AC886, AUClast | 5300 (1310)
  Oral (plasma): Quizartinib, AUCinf | 17600 (5500)
  Oral (plasma): AC886, AUCinf | 5580 (1200)

7. Secondary Outcome: Pharmacokinetic Parameter for Area Under the Plasma Concentration-Time Curve (AUC) Following Intravenous Administrations of Quizartinib
Description: Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0). Area under the concentration-time curve from the time of dosing to time (AUClast) and area under the concentration-time curve from the time of dosing extrapolated to infinity (AUCinf) were assessed for 14C-Quizartinib and 14C-AC886.
Time Frame: as for outcome 3
Population: Pharmacokinetic parameters were assessed in patients with available data in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | All Participants
Number analyzed (Participants) | 7
pg*h/mL
  Intravenous: 14C-Quizartinib, AUClast | 18800 (4950)
  Intravenous: 14C-AC886, AUClast | 5170 (1330)
  Intravenous: 14C-Quizartinib, AUCinf | 19600 (5390)
  Intravenous: 14C-AC886, AUCinf | 5620 (1270)

8. Secondary Outcome: Pharmacokinetic Parameter for Total Body Clearance (CL) Following Single-Dose Intravenous Administration of Quizartinib
Description: Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0). Total body clearance (CL) was assessed following single-dose IV administration for 14C-quizartinib.
Time Frame: as for outcome 3
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | All Participants
Number analyzed (Participants) | 8
L/h | 2.31 (0.624)

9. Secondary Outcome: Pharmacokinetic Parameter for Volume of Distribution (Vz) Following Following Single-Dose Intravenous Administration of Quizartinib
Description: Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0). Volume of distribution based on the terminal phase (Vz) was assessed following single-dose IV administration for 14C-quizartinib.
Time Frame: as for outcome 3
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | All Participants
Number analyzed (Participants) | 8
Liters | 318 (142)

10. Secondary Outcome: Pharmacokinetic Parameter of Metabolite to Parent Ratio (MPR) Based on Area Under the Curve Following Intravenous and Oral Administrations of Quizartinib
Description: Pharmacokinetic parameters were calculated using a non-compartmental approach. PK parameters were computed using Phoenix™ WinNonlin® (Version 8.0). MPR was assessed for AC886 and 14C-AC886.
Time Frame: Relative to oral dosing: Pre-dose (AC886 only), 1 hour (AC886 only), 2 hours (AC886 only), 4, 4.25, 4.5, 4.75, 5, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240, 288, 336, 384, 432, 480, and 504 hours
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable Population.
Measure: Mean (Standard Deviation); unit: metabolite-to-parent ratio
Arm/Group | All Participants
Number analyzed (Participants) | 8
metabolite-to-parent ratio
  Oral (plasma): MPR(AUClast), AC886 | 0.35 (0.164)
  Oral (plasma): MPR(AUCinf), AC886 | 0.35 (0.158)
  Intravenous: MPR(AUClast), 14C-AC886: number analyzed (Participants) | 7
  Intravenous: MPR(AUClast), 14C-AC886 | 0.29 (0.098)
  Intravenous: MPR(AUCinf), 14C-AC886 | 0.30 (0.093)

11. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event Following Intravenous and Oral Administrations of Quizartinib
Description: Treatment-emergent adverse events were coded using Medical Dictionary for Regulatory Activities (MedDRA) version 24.0.
Time Frame: Baseline up to approximately 6 weeks post-dose
Population: Treatment-emergent adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from baseline up to 6 weeks post-dose.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=8)
Cerumen impaction (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04796831/Prot_SAP_000.pdf